CLINICAL TRIAL: NCT04727671
Title: Effect of GnRH Agonist (Long Protocol) vs GnRH Antagonist (Flexible Protocol) on IVF/ICSI Outcomes in Polycystic Ovary Syndrome Patients.
Brief Title: Effect of GnRH Agonist vs GnRH Antagonist on IVF/ICSI Outcomes in Polycystic Ovary Syndrome Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ph-CT-4298
Record Dates: First submitted 2021-01-18; First posted 2021-01-27 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: In Vitro Fertilization; Intracytoplasmic Sperm Injection; Infertility; Polycystic Ovary Syndrome
Keywords: GnRH Agonist; GnRH Antagonist; Assisted reproduction technique; In Vitro Fertilization; Intracytoplasmic sperm injection; Polycystic Ovary Syndrome; Placental growth factor
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome | interventions — Triptorelin Pamoate; cetrorelix; Menotropins; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Agonist Group (Long protocol): (Active Comparator): The pituitary down-regulation in this group will be carried out using 0.05-0.1 mg of Triptorelin acetate subcutaneously (SC) once daily from the mid-luteal phase (day 21) of the menstrual cycle until the ovulation triggering day. When the suppressive effect is obtained, ovarian stimulation will commence with recombinant Follicle-Stimulating Hormone (r-FSH) or r-FSH + human Menopausal Gonadotropin (hMG) and the dose will be adjusted according to the ovarian response. Ovulation will be triggered by the administration of 10,000 IU of Human Chorionic Gonadotropin (hCG) when at least three follicles become more than 16-17 mm. After 35±2 hours of ovulation triggering, the oocytes will be retrieved by transvaginal ultrasound-guided follicle aspiration. Then they will be prepared to undergo an Intracytoplasmic Sperm Injection (ICSI).
  Interventions: Drug: Triptorelin acetate; Drug: recombinant-FSH or recombinant-FSH + human Menopausal Gonadotropin; Drug: Human Chorionic Gonadotropin (hCG)
- Antagonist Group (Flexible protocol): (Experimental): The ovarian stimulation in this group will be started with recombinant Follicle-Stimulating Hormone (r-FSH) or r-FSH + human Menopausal Gonadotropin (hMG) on the third day of the menstrual cycle and the dose will be adjusted according to the ovarian response. Initiation of 0.25 mg of GnRH antagonist; Cetrorelix; will take place after detecting a leading follicle diameter ≥ 14 mm. GnRH antagonist administration will be continued till the day of ovulation triggering, which will be accomplished by given 10,000 IU of Human Chorionic Gonadotropin (hCG) when at least three follicles become more than 16-17 mm. After 35±2 hours of ovulation triggering, the oocytes will be retrieved by transvaginal ultrasound-guided follicle aspiration. Then they will be prepared to undergo an Intracytoplasmic Sperm Injection (ICSI).
  Interventions: Drug: Cetrorelix; Drug: recombinant-FSH or recombinant-FSH + human Menopausal Gonadotropin; Drug: Human Chorionic Gonadotropin (hCG)

INTERVENTIONS:
Drug: Triptorelin acetate — 0.05-0.1 mg subcutaneously (SC) once daily from the mid-luteal phase (day 21) of the cycle until the day of ovulation triggering.
  Arms: Agonist Group (Long protocol):
Drug: Cetrorelix — 0.25 mg subcutaneously (SC) once daily starting from the day detecting a leading follicle diameter ≥ 14 mm until the day of ovulation triggering.
  Arms: Antagonist Group (Flexible protocol):
Drug: recombinant-FSH or recombinant-FSH + human Menopausal Gonadotropin — Dosage adjustment according to the ovarian response.
Drug: Human Chorionic Gonadotropin (hCG) — Ovulation will be triggered by the administration of 10,000 IU of Human Chorionic Gonadotropin (hCG) when at least three follicles become more than 16-17 mm.

SUMMARY:
This prospective, non-randomised, open-label, clinical trial is conducting on polycystic ovary syndrome (PCOS) subjects to compare the effects of two pituitary suppression regimens; GnRH Agonist-Long Protocol and GnRH Antagonist-Flexible Protocol on clinical and embryological IVF/ICSI outcomes, and on the follicular fluid levels of Placental Growth Factor (PlGF); which is known for his pivotal role in the regulation of ovulation, embryo development, and implantation

ELIGIBILITY:
Inclusion Criteria:

* PCOS women diagnosed according to the Rotterdam criteria undergoing IVF/ICSI.
* Age: 18-39 years.
* Both ovaries present.

Exclusion Criteria:

* Age ≥ 40 years.
* History of three or more previous IVF failures.
* Patients with hormonal disorders like hyperprolactinemia, thyroid disorders.
* Patients who previously undergo Unilateral Oophorectomy.
* Patients with chronic diseases: diabetes mellitus, cardiovascular diseases, liver diseases, kidney diseases.
* Patients with diseases may affect IVF outcomes: Endometriosis, uterine fibroids, Hydrosalpinx, Adenomyosis, autoimmune diseases,
* Cancer.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-12-22 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Follicular fluid Placental Growth Factor (PlGF) Concentrations: | Immediately after oocyte retrieval (35±2 hours after hCG administration)
  Follicular fluid samples will be obtained on the day of oocyte retrieval, then they will be centrifuged to eliminate cellular elements and debris. After that, the supernatants will be frozen at -80 until assayed using an Elisa kit.

SECONDARY OUTCOMES:
Number of oocytes retrieved | Immediately after oocyte retrieval (35±2 hours after hCG administration)
  The oocytes will be retrieved by transvaginal ultrasound-guided follicle aspiration 35±2 hours after hCG administration.
Number of Metaphase II Oocytes (MII): | Within two hours after oocyte retrieval
  The oocyte maturity will be assessed using Nikon SMZ1500 stereoscope.
Maturation Rate%: | Within two hours after oocyte retrieval
  Maturation Rate is calculated by dividing the number of mature (MII) oocytes by the number of retrieved oocytes.
Fertilization Rate%: | 16-18 hours after microinjection.
  Fertilization Rate is calculated by dividing the number of obtained zygote (2PN) by the number of injected oocytes.
Cleavage Rate%: | Day 2 after microinjection.
  Cleavage rate is calculated by dividing the number of cleavaged embryos by the number of zygotes (2PN).
Embryo Quality: | Day of transfer (2 or 3 days after microinjection).
  Embryos are assessed using Nikon SMZ1500 stereoscope based on ESHRE criteria (2011).
High Quality Embryos rate%: | Day of transfer (2 or 3 days after microinjection).
  High Quality Embryos rate is calculated by dividing the number of high quality embryos (Grade I) by the total number of cleavaged embryos.
Biochemical Pregnancy Rate% (Per Embryo Transfer): | 2 weeks after embryo transfer
  Biochemical pregnancy is defined as a positive serum beta-hCG pregnancy test after 2 weeks of embryo transfer. The biochemical pregnancy rate is calculated by dividing the number of women who are biochemically pregnant by the number of women who have at least 1 embryo transferred.
Clinical Pregnancy Rate% (Per Embryo Transfer): | 3-4 weeks after embryo transfer
  Clinical pregnancy is defined as the presence of a gestational sac on ultrasound after 3-4 weeks of embryo transfer. The clinical pregnancy rate is calculated as by dividing the number of women who are clinically pregnant divided by the number of women who have at least 1 embryo transferred.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Kadoura, B Pharm, MD, Principal Investigator — Department of Pharmaceutics and Pharmaceutical Technology, Faculty of Pharmacy, Damascus University, Damascus, Syria; Abdul Hakim Nattouf, MD, PhD, Study Director — Professor at Department of Pharmaceutics and Pharmaceutical Technology, Faculty of Pharmacy, Damascus University, Damascus, Syria; Marwan Alhalabi, MD, PhD, Study Director — Professor at Department of Embryology and Reproductive Medicine, Faculty of Medicine, Damascus University, Damascus, Syria.
Locations (1):
- Orient Hospital, Damascus, Syria

REFERENCES:
- [Background] Azziz R, Carmina E, Chen Z, Dunaif A, Laven JS, Legro RS, Lizneva D, Natterson-Horowtiz B, Teede HJ, Yildiz BO. Polycystic ovary syndrome. Nat Rev Dis Primers. 2016 Aug 11;2:16057. doi: 10.1038/nrdp.2016.57. PMID 27510637
- [Background] Dennett CC, Simon J. The role of polycystic ovary syndrome in reproductive and metabolic health: overview and approaches for treatment. Diabetes Spectr. 2015 May;28(2):116-20. doi: 10.2337/diaspect.28.2.116. No abstract available. PMID 25987810
- [Background] Lai Q, Zhang H, Zhu G, Li Y, Jin L, He L, Zhang Z, Yang P, Yu Q, Zhang S, Xu JF, Wang CY. Comparison of the GnRH agonist and antagonist protocol on the same patients in assisted reproduction during controlled ovarian stimulation cycles. Int J Clin Exp Pathol. 2013 Aug 15;6(9):1903-10. eCollection 2013. PMID 24040457
- [Background] Hoseini FS, Noori Mugahi SM, Akbari-Asbagh F, Eftekhari-Yazdi P, Aflatoonian B, Aghaee-Bakhtiari SH, Aflatoonian R, Salsabili N. A randomized controlled trial of gonadotropin-releasing hormone agonist versus gonadotropin-releasing hormone antagonist in Iranian infertile couples: oocyte gene expression. Daru. 2014 Oct 7;22(1):67. doi: 10.1186/s40199-014-0067-4. PMID 25288473
- [Background] Al-Inany HG, Youssef MA, Ayeleke RO, Brown J, Lam WS, Broekmans FJ. Gonadotrophin-releasing hormone antagonists for assisted reproductive technology. Cochrane Database Syst Rev. 2016 Apr 29;4(4):CD001750. doi: 10.1002/14651858.CD001750.pub4. PMID 27126581
- [Background] Binder NK, Evans J, Salamonsen LA, Gardner DK, Kaitu'u-Lino TJ, Hannan NJ. Placental Growth Factor Is Secreted by the Human Endometrium and Has Potential Important Functions during Embryo Development and Implantation. PLoS One. 2016 Oct 6;11(10):e0163096. doi: 10.1371/journal.pone.0163096. eCollection 2016. PMID 27711226
- [Background] Bender HR, Trau HA, Duffy DM. Placental Growth Factor Is Required for Ovulation, Luteinization, and Angiogenesis in Primate Ovulatory Follicles. Endocrinology. 2018 Feb 1;159(2):710-722. doi: 10.1210/en.2017-00739. PMID 29095972
- [Background] Tal R, Seifer DB, Grazi RV, Malter HE. Follicular fluid placental growth factor is increased in polycystic ovarian syndrome: correlation with ovarian stimulation. Reprod Biol Endocrinol. 2014 Aug 20;12:82. doi: 10.1186/1477-7827-12-82. PMID 25141961
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538
- [Background] Alpha Scientists in Reproductive Medicine and ESHRE Special Interest Group of Embryology. The Istanbul consensus workshop on embryo assessment: proceedings of an expert meeting. Hum Reprod. 2011 Jun;26(6):1270-83. doi: 10.1093/humrep/der037. Epub 2011 Apr 18. PMID 21502182